CLINICAL TRIAL: NCT02608086
Title: Psychological First Aid: A Randomized-controlled Trial of Adults Affected by Non-intentional Trauma in the Emergency Room
Brief Title: Psychological First Aid (PFA): RCT Adults Non-intentional Trauma Emergency Room
Acronym: PFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 15-196; FONDAP 15110017/2011 (Other Grant/Funding Number: CIGIDEN)
Record Dates: First submitted 2015-11-03; First posted 2015-11-18 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: PTSD
Keywords: PTSD; Trauma; Emergency; RCT; Psychological First Aid
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries; Emergencies | interventions — Psychological First Aid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Other): Flyer "What can I do facing a crisis?"
  Interventions: Behavioral: Psychoeducation
- Psychological First Aid (Experimental): Psychological First Aid according to an adapted protocol based on the WHO PFA Operation Guide 2012 Brochure "Network and Services" Flyer "What can I do facing a crisis?".
  Interventions: Behavioral: Psychological First Aid

INTERVENTIONS:
Behavioral: Psychoeducation — Participants in Control Group will be delivered a flyer named "What can I do facing a crisis?", containing information about normal reactions to crisis, what to do to return to normal life and which are the signals of an initial trauma.
  Arms: Control
Behavioral: Psychological First Aid — Psychology students (PFA Providers) will intervene according to an adapted protocol based on the WHO PFA Operation Guide 2012. Protocol for this study contemplates 4 steps: 1. Active Listening 2. Relaxing and Breathing Techniques 3. Help in prioritizing needs 4. Help in contacting network and services. Moreover, participants in this group will receive a brochure with full contact information of public network, and a flyer named "What can I do facing a crisis?".
  Other Names: PFA
  Arms: Psychological First Aid

SUMMARY:
Psychological First Aid (PFA) is currently the most recommended early intervention for people affected by recent traumatic events, especially in the aftermath of natural disasters. Unfortunately, there is no evidence that PFA neither prevents Post-Traumatic Stress Disorder (PTSD) nor other post-traumatic disorders or symptoms of distress. This project aims to evaluate the efficacy and safety of Psychological First Aid for the prevention of PTSD and other post-traumatic disorders or symptoms.

DETAILED DESCRIPTION:
Background: Psychological First Aid (PFA) is currently the most recommended early intervention for people affected by recent traumatic events, especially in the aftermath of natural disasters. Unfortunately, there is no evidence that PFA neither prevents Post-Traumatic Stress Disorder (PTSD) nor other post-traumatic disorders or symptoms of distress.

Objective: This project aims to evaluate the efficacy and safety of Psychological First Aid for the prevention of PTSD and other post-traumatic disorders and/or symptoms.

Population: Investigators will perform a 1:1 randomized-controlled trial of 200 adults recently affected (<=72 hours) by a non-intentional trauma who consult to the emergency room of a public hospital. Investigators estimated a sample size of 200 individuals in order to detect a 50% Relative Risk Reduction (RRR), with a power of 80%, a statistical significance (alpha) of 5% and 34,4% of PTSD prevalence in the control group, what is consistent with prevalences observed in a similar sample by Fullerton, Ursano, Epstein, Crowley, Vance et al. (2001).

Intervention: In the emergency room, undergraduate psychology students, previously trained and certified in PFA, will search and randomize suitable patients to either PFA or treatment as usual (TAU). They will provide PFA according to a protocol based on the WHO PFA Operation Guide to those patients included in the active group. Everyone correctly randomized will be followed and clinically evaluated one month after the intervention (endpoint).

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years old) concurring to the emergency room, either as a patient himself or companion, who have been victims of a recent unintentional trauma (less than 72 hours ago), and meet one of the following criteria:
* Direct victim, as a family or as a witness, of a situation that was or is currently life threatening.
* Direct victim, as a family or as a witness, of a situation that affected or currently seriously endangers the physical integrity.

For example, such situations include serious accidents, catastrophic illness, highly painful medical procedures, bad medical news, natural disasters, fires, witnessing another person violent death, explosions, among others.

Exclusion Criteria:

* Does not understand Spanish
* Child and adolescent (< 18 years old)
* Can not remember traumatic experience recently experienced
* Psychosis (loss of reality testing)
* People in life-threatening or health instability situation, requiring equipment for life support incompatible with this application protocol (serious fractures, severe bleeding wounds with uncontrolled excruciating pain, unstable myocardial infarction, etc.). Will be the attending physician whom inform the patient if this exclusion criterion is met.
* Relatives of people in imminent life-threatening or recently died in the emergency room where the offer to participate in the research can cause even greater discomfort.
* Impairment of consciousness (Glasgow < 15)
* Intoxication
* Loss of consciousness for more than 5 minutes.
* Direct and indirect victims of intentional trauma (eg. assault, kidnapping, sexual abuse, terrorist attack, etc).
* Patients being treated for a psychiatric disorder diagnosed by a doctor (personality disorder is excluded) (eg. schizophrenia, mental retardation, autism, obsessive compulsive disorder, bipolar disorder, depression, Alzheimer's disease, panic disorder, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2015-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
PTSD Prevalence | 1 month
  PTSD prevalence according to Composite International Diagnostic Interview (CIDI)

SECONDARY OUTCOMES:
PTSD symptoms | 1 month
  According to the PCL-C

OTHER OUTCOMES:
Self-reported depressive symptoms | 1 month
  According to Beck Depression Inventory
Perceived Social Support | 1 month
  According to Multidimensional Scale of Perceived Social Support (MSPSS)
Satisfaction with Intervention | Once intervention has finished, an estimate time frame of 90 minutes for "active group" or 50 minutes for "control group"
  According to Analog Visual Scale
Peri-traumatic dissociative experiences | 1 month
  According to PDEQ
Peri-traumatic Distress | 1 month
  According to Peri-traumatic Distress Inventory (PDI)
Previous traumatic experiences | 1 month
  According to TQ

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo A. Figueroa, MD, Principal Investigator — CIGIDEN
Locations (5):
- Chile (5):
  - Hospital Barros Luco Trudeau, Santiago, Santiago Metropolitan
  - Hospital Clínico UC, Santiago, Santiago Metropolitan
  - Hospital del Trabajador, Santiago, Santiago Metropolitan
  - Hospital Dr. Sótero del Río, Santiago, Santiago Metropolitan
  - Hospital Padre Hurtado, Santiago, Santiago Metropolitan

REFERENCES:
- [Background] Breslau N. The epidemiology of posttraumatic stress disorder: what is the extent of the problem? J Clin Psychiatry. 2001;62 Suppl 17:16-22. PMID 11495091
- [Background] Carlson EB, Smith SR, Palmieri PA, Dalenberg C, Ruzek JI, Kimerling R, Burling TA, Spain DA. Development and validation of a brief self-report measure of trauma exposure: the Trauma History Screen. Psychol Assess. 2011 Jun;23(2):463-77. doi: 10.1037/a0022294. PMID 21517189
- [Background] Everly GS Jr, Mitchell JT. The debriefing "controversy" and crisis intervention: a review of lexical and substantive issues. Int J Emerg Ment Health. 2000 Fall;2(4):211-25. PMID 11217152
- [Background] Flannery RB Jr, Everly GS Jr. Crisis intervention: a review. Int J Emerg Ment Health. 2000 Spring;2(2):119-25. PMID 11232174
- [Background] Friedman MJ, Resick PA, Bryant RA, Brewin CR. Considering PTSD for DSM-5. Depress Anxiety. 2011 Sep;28(9):750-69. doi: 10.1002/da.20767. Epub 2010 Dec 13. PMID 21910184
- [Background] Green BL, Lindy JD, Grace MC, Leonard AC. Chronic posttraumatic stress disorder and diagnostic comorbidity in a disaster sample. J Nerv Ment Dis. 1992 Dec;180(12):760-6. doi: 10.1097/00005053-199212000-00004. PMID 1469374
- [Background] Hobfoll SE, Watson P, Bell CC, Bryant RA, Brymer MJ, Friedman MJ, Friedman M, Gersons BP, de Jong JT, Layne CM, Maguen S, Neria Y, Norwood AE, Pynoos RS, Reissman D, Ruzek JI, Shalev AY, Solomon Z, Steinberg AM, Ursano RJ. Five essential elements of immediate and mid-term mass trauma intervention: empirical evidence. Psychiatry. 2007 Winter;70(4):283-315; discussion 316-69. doi: 10.1521/psyc.2007.70.4.283. PMID 18181708
- [Background] Hoge EA, Worthington JJ, Nagurney JT, Chang Y, Kay EB, Feterowski CM, Katzman AR, Goetz JM, Rosasco ML, Lasko NB, Zusman RM, Pollack MH, Orr SP, Pitman RK. Effect of acute posttrauma propranolol on PTSD outcome and physiological responses during script-driven imagery. CNS Neurosci Ther. 2012 Jan;18(1):21-7. doi: 10.1111/j.1755-5949.2010.00227.x. Epub 2011 Jan 10. PMID 22070357
- [Background] Kessler RC. Posttraumatic stress disorder: the burden to the individual and to society. J Clin Psychiatry. 2000;61 Suppl 5:4-12; discussion 13-4. PMID 10761674
- [Background] Kessler RC, Sonnega A, Bromet E, Hughes M, Nelson CB. Posttraumatic stress disorder in the National Comorbidity Survey. Arch Gen Psychiatry. 1995 Dec;52(12):1048-60. doi: 10.1001/archpsyc.1995.03950240066012. PMID 7492257
- [Background] Norris FH, Murphy AD, Baker CK, Perilla JL, Rodriguez FG, Rodriguez Jde J. Epidemiology of trauma and posttraumatic stress disorder in Mexico. J Abnorm Psychol. 2003 Nov;112(4):646-56. doi: 10.1037/0021-843X.112.4.646. PMID 14674876
- [Background] Ozer EJ, Best SR, Lipsey TL, Weiss DS. Predictors of posttraumatic stress disorder and symptoms in adults: a meta-analysis. Psychol Bull. 2003 Jan;129(1):52-73. doi: 10.1037/0033-2909.129.1.52. PMID 12555794
- [Background] Perkonigg A, Kessler RC, Storz S, Wittchen H -U. Traumatic events and post-traumatic stress disorder in the community: prevalence, risk factors and comorbidity. Acta Psychiatr Scand. 2000 Jan;101(1):46-59. doi: 10.1034/j.1600-0447.2000.101001046.x. PMID 10674950
- [Background] Ramos-Brieva JA, Cordero Villafafila A. [Validation of the Castillian version of the Hamilton Rating Scale for Depression]. Actas Luso Esp Neurol Psiquiatr Cienc Afines. 1986 Jul-Aug;14(4):324-34. No abstract available. Spanish. PMID 3776732
- [Background] Rose S, Bisson J, Churchill R, Wessely S. Psychological debriefing for preventing post traumatic stress disorder (PTSD). Cochrane Database Syst Rev. 2002;(2):CD000560. doi: 10.1002/14651858.CD000560. PMID 12076399
- [Background] Rothbaum BO, Kearns MC, Price M, Malcoun E, Davis M, Ressler KJ, Lang D, Houry D. Early intervention may prevent the development of posttraumatic stress disorder: a randomized pilot civilian study with modified prolonged exposure. Biol Psychiatry. 2012 Dec 1;72(11):957-63. doi: 10.1016/j.biopsych.2012.06.002. Epub 2012 Jul 4. PMID 22766415
- [Background] Schelling G, Roozendaal B, Krauseneck T, Schmoelz M, DE Quervain D, Briegel J. Efficacy of hydrocortisone in preventing posttraumatic stress disorder following critical illness and major surgery. Ann N Y Acad Sci. 2006 Jul;1071:46-53. doi: 10.1196/annals.1364.005. PMID 16891561
- [Background] Stein MB, McQuaid JR, Pedrelli P, Lenox R, McCahill ME. Posttraumatic stress disorder in the primary care medical setting. Gen Hosp Psychiatry. 2000 Jul-Aug;22(4):261-9. doi: 10.1016/s0163-8343(00)00080-3. PMID 10936633
- [Background] Teasdale G, Jennett B. Assessment of coma and impaired consciousness. A practical scale. Lancet. 1974 Jul 13;2(7872):81-4. doi: 10.1016/s0140-6736(74)91639-0. No abstract available. PMID 4136544
- [Background] Vera-Villarroel P, Zych I, Celis-Atenas K, Cordova-Rubio N, Buela-Casal G. Chilean validation of the Posttraumatic Stress Disorder Checklist-Civilian version (PCL-C) after the earthquake on February 27, 2010. Psychol Rep. 2011 Aug;109(1):47-58. doi: 10.2466/02.13.15.17.PR0.109.4.47-58. PMID 22049647
- [Background] Vicente B, Kohn R, Rioseco P, Saldivia S, Levav I, Torres S. Lifetime and 12-month prevalence of DSM-III-R disorders in the Chile psychiatric prevalence study. Am J Psychiatry. 2006 Aug;163(8):1362-70. doi: 10.1176/ajp.2006.163.8.1362. PMID 16877648
- [Background] Watson PJ, Brymer MJ, Bonanno GA. Postdisaster psychological intervention since 9/11. Am Psychol. 2011 Sep;66(6):482-94. doi: 10.1037/a0024806. PMID 21823776
- [Background] Zlotnick C, Johnson J, Kohn R, Vicente B, Rioseco P, Saldivia S. Epidemiology of trauma, post-traumatic stress disorder (PTSD) and co-morbid disorders in Chile. Psychol Med. 2006 Nov;36(11):1523-33. doi: 10.1017/S0033291706008282. Epub 2006 Jul 20. PMID 16854253
- [Background] Dieltjens T, Moonens I, Van Praet K, De Buck E, Vandekerckhove P. A systematic literature search on psychological first aid: lack of evidence to develop guidelines. PLoS One. 2014 Dec 12;9(12):e114714. doi: 10.1371/journal.pone.0114714. eCollection 2014. PMID 25503520
- See also: CIGIDEN website — http://www.cigiden.cl
- See also: Related Info — http://www.info-trauma.org